CLINICAL TRIAL: NCT03855553
Title: Disseminating Eating Disorders Education and Treatment Across Multiple Levels of Care: Improving Access in the Rhode Island Medicaid Population
Brief Title: Project CORE: Disseminating Eating Disorders Treatment
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1319865
Record Dates: First submitted 2019-02-21; First posted 2019-02-26 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2020-08

CONDITIONS: Anorexia Nervosa/Bulimia; Anorexia Nervosa Restricting Type; Eating Disorders in Adolescence
Keywords: Anorexia Nervosa; Bulimia Nervosa; Eating Disorders; Adolescence; Clinical Training; Community Outreach; Family Based Treatment; Enhanced Cognitive Behavioral Therapy
MeSH Terms: conditions — Anorexia Nervosa; Bulimia; Bulimia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FBT (Experimental): 10 families will be randomized to receive 10 - 16 weeks of eating disorder treatment for their adolescent.
  Interventions: Behavioral: Family Based Treatment
- CBT-E (Experimental): 10 families will be randomized to receive 10 - 16 weeks of eating disorder treatment for their adolescent.
  Interventions: Behavioral: Enhanced Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Family Based Treatment — 10 families will be randomized to receive 10 - 16 weeks of Family Based Treatment (FBT), the "gold standard" in eating disorder treatment for adolescents. FBT is a highly structured behavioral intervention in which caregivers are charged with the primary task of re-feeding their child and normalizing his or her eating behaviors and weight status.
  Other Names: FBT
  Arms: FBT
Behavioral: Enhanced Cognitive Behavioral Therapy — 10 families will be randomized to receive 10 - 16 weeks of Enhanced Cognitive Behavioral Therapy (CBT-E), a clinically validated treatment for adolescent eating disorders. CBT-E is a short-term, individual treatment focused on normalizing eating behaviors and modifying underlying cognitions that contribute to the maintenance of eating disorder behaviors (e.g., over-importance of shape and weight in one's self-evaluation).
  Other Names: CBT-E
  Arms: CBT-E

SUMMARY:
The goals of this project are to 1) develop training opportunities for master's-level and pre-doctoral psychology students in evidence-based assessment and treatment of adolescent EDs; 2) to provide the healthcare workforce, including licensed health professionals such as primary care physicians and behavioral health interventionists, with knowledge and competence to recognize early symptoms of and intervention strategies for EDs; and 3) to test the efficacy of delivering two evidence-based treatments for adolescent eating disorders, Family Based Treatment (FBT) and Enhanced Cognitive Behavioral Therapy (CBT-E), in the home-based setting.

DETAILED DESCRIPTION:
The complete project will incorporate three phases. Phase I is designed to gather information from existing licensed health professionals in the community who serve Medicaid populations on their knowledge needs and priorities related to screening and intervening with patients with eating disorders. Phase I will comprise eating disorder psycho-education, implementation of workshops, and supervision among primary care professionals and mental health workers. Responses will inform the content of in-services and program development (e.g., monthly consultation services, ongoing multi-family support groups) provided in Phase II.

During Phase II, families containing a child with a restrictive-type eating disorder will be recruited to receive treatment from the clinicians assessed and trained during Phase I. Families will be assigned to receive either Family Based Treatment (FBT) or Enhanced Cognitive Behavioral Therapy (CBT-E) to treat their adolescent's eating disorder. Treatment will occur over 10-16 weeks, depending on the family's needs and availability. Families will be assessed at pre-treatment, post-treatment, and 1-year follow-up.

Phase III will consist of follow-up with the families and clinicians, and further development of training/education approaches for the Rhode Island healthcare workforce.

ELIGIBILITY:
Inclusion criteria include:

* meets criteria for AN, atypical AN, or BN according to DSM-5 diagnostic criteria
* is currently living at home
* is medically stable for outpatient treatment according to the recommended thresholds of the American Academy of Pediatrics and the Society of Adolescent Medicine (e.g., ≥75% of expected body weight, heartrate ≥50 beats per minute)
* if on a psychotropic medication, meets all eligibility criteria while on stable dose of psychotropic medication (8 weeks) for a co-morbid condition
* speaks English
* be available for long-term follow-up.

Exclusion criteria include:

* associated physical illness that necessitates hospitalization
* psychotic illness/other mental illness requiring hospitalization
* current dependence on drugs or alcohol
* physical conditions (e.g. diabetes mellitus, pregnancy) known to influence eating or weight
* concurrent involvement in other psychological treatment for an eating disorder
* developmental delay that would preclude participation in the intervention.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
BMI percentile | post treatment (week 17)
BMI percentile | 1 year follow up
Eating disorder symptomology, as assessed by the EDE-Q. | post treatment (week 17)
  Patient will complete the Eating Disorder Examination Questionnaire (EDE-Q) to assess the frequency and severity of specific eating disorder behaviors and cognitions. Averages of the 28-item measure range from 0 to 6, with higher score indicating higher eating disorder symptomology.
Eating disorder symptomology, as assessed by the ED-15. | post treatment (week 17)
  Patient will complete the Eating Disorder 15 (ED-15) to assess the frequency and severity of specific eating disorder behaviors and cognitions. Average scores from the 15-item measure range from 1 - 5, with higher scores indicating higher eating disorder symptomology.
Eating disorder symptomology, as assessed by EDE-Q | 1 year follow-up
  Patient will complete the Eating Disorder Examination Questionnaire (EDE-Q) to assess the frequency and severity of specific eating disorder behaviors and cognitions. Average scores of the 28-item measure range from 0 to 6, with higher score indicating higher eating disorder symptomology.
Eating disorder symptomology, as assessed by ED-15. | 1 year follow-up
  Patient will complete the Eating Disorder 15 (ED-15) to assess the frequency and severity of specific eating disorder behaviors and cognitions. Average scores from the 15-item measure range from 1 - 5, with higher scores indicating higher eating disorder symptomology.
Perceived efficacy of treatment, as assessed by the TSPE | post treatment (week 17)
  One item from the Treatment Suitability and Patient Expectancy (TSPE) survey will assess how successful the patient perceived treatment to be. This item ranges from 0 - 10, with higher scores indicating higher perceived efficacy.
Perceived efficacy of treatment, as assessed by the CSQ | post treatment (week 17)
  The Client Satisfaction Questionnaire (CSQ) is an 8-item measure that assesses how successful the patient perceived treatment to be. Average scores range from 1 - 4, with higher scores indicating higher satisfaction and perceived efficacy.
Perceived efficacy of treatment, as assessed by the CSQ | 1 year follow-up
  The Client Satisfaction Questionnaire (CSQ) is an 8-item measure that assesses how successful the patient perceived treatment to be. Average scores range from 1 - 4, with higher scores indicating higher satisfaction and perceived efficacy.
Perceived efficacy of treatment, as assessed by the TSPE. | 1 year follow-up
  One item from the Treatment Suitability and Patient Expectancy (TSPE) survey will assess how successful the patient perceived treatment to be. This item ranges from 0 - 10, with higher scores indicating higher perceived efficacy.
Perceived feasibility of treatment, as assessed by the TSPE. | post treatment (week 17)
  One item from the Treatment Suitability and Patient Expectancy (TSPE) survey will assess how feasible the patient perceived treatment to be. This item ranges from 0 - 10, with higher scores indicating higher feasibility.
Perceived feasibility of treatment, as assessed by the CSQ. | post treatment (week 17)
  Two items from the 8-item Client Satisfaction Questionnaire (CSQ) will assess how suitable/feasible treatment was based on the patient's needs, family dynamics, schedule constraints, etc. Average scores range from 1 - 4, with higher scores indicating higher feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea B. Goldschmidt, Ph.D., Principal Investigator — Weight Control & Diabetes Research Center; Christina Tortolani, Ph.D., Principal Investigator — Rhode Island College
Locations (1):
- The Weight Control & Diabetes Research Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No